CLINICAL TRIAL: NCT04769050
Title: A Phase II, Single-center, Dynamic Observational Study With PET of 68Ga-HER2-affibody in Anti-HER2 Treatment
Brief Title: Dynamic Observational Study With PET of 68Ga-HER2-affibody in Anti-HER2 Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Director of department of medical oncology, Fudan University
Other Study IDs: DOLPHIN
Record Dates: First submitted 2021-02-15; First posted 2021-02-24 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ado-Trastuzumab Emtansine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First-line patients: First-line treatment of HER2-positive metastatic breast cancer patients
  Interventions: Drug: Docetaxel combined with Trastuzumab±Pertuzumab
- Second-line patients: Second-line treatment of HER2-positive metastatic breast cancer patients
  Interventions: Drug: T-DM1 or Capecitabine combined with Pyrotinib regimen.

INTERVENTIONS:
Drug: Docetaxel combined with Trastuzumab±Pertuzumab — Docetaxel, 75 mg/m2 ivgtt d1 q3w Trastuzumab, 6 mg/kg(8 mg/kg for initial dose) ivgtt d1 q3w Pertuzumab, 420mg(840mg for initial dose) ivgtt d1 q3w
  Groups: First-line patients
Drug: T-DM1 or Capecitabine combined with Pyrotinib regimen. — T-DM1, 3.6mg/kg(8 mg/kg for initial dose) ivgtt d1 q3w Capecitabine, 1250 mg/m2 bid po d1-14 q3w Pyrotinib, 400mg po daily (continuously)
  Groups: Second-line patients

SUMMARY:
Dynamic observationaL study with PET of 68Ga-HER2-affibody in anti-HER2 treatment

DETAILED DESCRIPTION:
Participants participated in the screening period visit, and received HER2-PET and 18 F-FDG PET/CT examinations before receiving tumor treatment, after receiving 2 cycles of chemotherapy, and after disease progression. Patients of first-line received docetaxel combined with trastuzumab±pertuzumab regimen, and patients of second-line received T-DM1 monotherapy or capecitabine combined with pyrrotinib regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily joined the study, signed informed consent, and had good compliance.
2. Female patients aged over 18 years (including cutoff value).
3. an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
4. Patients with HER2 positive recurrent or metastatic breast cancer confirmed by histopathology.
5. At least one extracranial measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1.
6. Previously received no more than 1 prior lines of systemic chemotherapy for metastatic breast cancer
7. Life expectancy ≥ 12 weeks.
8. Adequate function of major organs meets the following requirements (no blood components and cell growth factors have been used within 14 days before randomization):

   * Neutrophils ≥ 1.5×10^9/L
   * Platelets ≥ 75×10^9/L
   * Hemoglobin ≥ 80g/L
   * Total bilirubin≤ 1.5 × the upper limit of normal (ULN)
   * ALT and AST ≤ 3 × ULN
   * BUN and Cr ≤ 1.5 × ULN
   * Left ventricular ejection fraction (LVEF) ≥ 50%
   * QTcF(Fridericia correction) ≤ 470 ms

Exclusion Criteria:

1. The subject has untreated central nervous system (CNS) metastases.
2. Patients who have undergone systemic, radical brain or meningeal metastasis (radiotherapy or surgery), but have been confirmed to have been stable for at least 4 weeks, and who have stopped systemic hormonal therapy for more than 2 weeks without clinical symptoms can be included.
3. Received systemic therapy such as chemotherapy, molecular targeted therapyment;received endocrine therapy within 2 weeks before enrollment.
4. Patients with other malignant tumors within 3 years or at the sametime(except for cured skin basal cell carcinoma and cervical carcinomain situ).
5. Have undergone major surgical procedures or significant trauma within 4 weeks prior to randomization, or are expected to undergo major surgery.
6. Pregnant women, lactating female, or women of childbearing age who are unwilling to take effective contraceptive measures.
7. Have a history of allergies to the drug components of this regimen.
8. Patients with active HBV and HCV infection; stable hepatitis B after drug treatment (HBV virus copy number is higher than the upper limit of reference value) and cured hepatitis C patients (HCV virus copy number exceeds the lower limit of detection method).
9. History of immunodeficiency, including HIV positive, or other acquired or congenital immunodeficiency disease, history of organ transplantation.
10. History of cardiac dysfunction, include(1)angina (2)clinical significant arrythmia or require drug intervention (3)myocardial infarction (4)heart failure (5) other cardiac dysfunction (judged by the physician); any cardiac or nephric abnormal ≥ grade 2 found in screening.
11. Female patients who are pregnancy, lactation or women who are ofchildbearing potential tested positive in baseline pregnancy test.
12. Childbearing female who refuse to accept any contraception practice.
13. Determined by the physician, any serious coexisting disease might be harmful to the patient's safety or avoid the patients from accomplishing the treatment(e.g serious hypertension, diabetes, thyroid dysfunction,active infection etc.).
14. History of neurological or psychiatric disorders, including epilepsy or dementia.
15. Severe infections within 4 weeks prior to first dose (eg, intravenous infusion of antibiotics, antifungal or antiviral drugs according to clinical protocols), or unexplained fever (T > 38.3 °C ) during screening or prior to first administration

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with HER2 positive recurrent or metastatic breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-02-18 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The correlation between the change of HER2-PET at baseline and after 2 courses of treatment and ORR. | 2 year
  The correlation between the percent change in standardized uptake value (SUV) on 68Ga-Affibody HER-2 Imaging PET at baseline and after 2 courses of treatment and objective response rate(ORR).

SECONDARY OUTCOMES:
The correlation between the change of HER2-PET at baseline and after 2 courses of treatment and PFS | 2 year
  The correlation between the percent change in SUV on 68Ga-Affibody HER-2 Imaging PET at baseline and after 2 courses of treatment and progression-free survival(PFS).
The correlation between baseline HER2 expression and ORR, PFS | 2 year
  The correlation between the baseline SUVmax on 68Ga-Affibody HER-2 Imaging PET and ORR, PFS.
The correlation between heterogeneity of baseline HER2 expression and ORR, PFS | 2 year
  The correlation between heterogeneity of the baseline SUVmax on 68Ga-Affibody HER-2 Imaging PET and ORR, PFS.
To explore the condition of HER2-PET when PD. | 2 year
  To detection the change in SUVmax on 68Ga-Affibody HER-2 Imaging PET when progressive disease(PD).

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, MD, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No